CLINICAL TRIAL: NCT00959686
Title: Bendamustine in Patients With Refractory or Relapsed T-cell Lymphoma. A Phase II Multicenter Study "BENTLY"
Brief Title: Bendamustine in Patients With Refractory or Relapsed T-cell Lymphoma
Acronym: BENTLY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Mundipharma Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: "BENTLY"
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2011-06

CONDITIONS: T-cell Lymphoma
Keywords: Bendamustine refractory or relapsed T-cell lymphoma.
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine (Experimental): Bendamustine at the dose of 120 mg/m2 IV over 60 minutes on days 1 and 2 every 21 days for 6 cycles
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — Bendamustine at the dose of 120 mg/m2 IV over 60 minutes on days 1 and 2 every 21 days for 6 cycles
  Other Names: Ribomustin®

SUMMARY:
A Phase II clinical study to determine the efficacy of single agent Bendamustine for T cell lymphoma "BENTLY".

DETAILED DESCRIPTION:
The primary objective of this study is to define the activity of Bendamustine for the treatment of T cells lymphomas. The activity of Bendamustine is determined by the response rate (RR) to the treatment within 22 days after intravenous infusion which enables to get a confidence interval of 95 % for the probability of an overall response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years.
* Refractory or relapsed peripheral T-cell NHL (PTCL)
* Cutaneous T cell lymphoma (CTCL) in relapse or refractory to topical therapy
* ECOG score less than 2
* No major organ dysfunction unrelated to lymphoma.

Exclusion Criteria:

* Pregnant or breast feeding women
* ECOG score > 2
* Estimate survival time < 3 months
* Active infection or severe organ dysfunction or psychiatric condition that unable patients to receive chemotherapy
* Creatinine clearance < 10 ml/min or severe hepatic dysfunction not related to lymphoma.
* Previous chemotherapy/immunotherapy within 3 weeks before study entry
* Known seropositive for or active viral infection HIV, EBV, HCV
* CNS lymphoma
* T-cell Leukemia lymphoma associated with HTLV1
* Sezary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Determine the overall response rate (ORR) (CR+CRu+PR) | 36 months follow-up

SECONDARY OUTCOMES:
Evaluation of the tolerance and Safety of bendamustine in this subset of patients | 36 months follow-up
Determination of the progression free survival (PFS), time to treatment failure (TTF), time to progression (TTP), overall survival (OS) and the duration of response. | 36 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Gandhi DAMAJ, MD MS, Principal Investigator — French Innovative Leukemia Organisation; Rémy GRESSIN, MD MS, Principal Investigator — French Innovative Leukemia Organisation; THierry LAMY, PD MS, Principal Investigator — French Innovative Leukemia Organisation; Olivier TOURNILHAC, PD MS, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Dr Gandhi DAMAJ, Amiens, France

REFERENCES:
- [Derived] Damaj G, Gressin R, Bouabdallah K, Cartron G, Choufi B, Gyan E, Banos A, Jaccard A, Park S, Tournilhac O, Schiano-de Collela JM, Voillat L, Joly B, Le Gouill S, Saad A, Cony-Makhoul P, Vilque JP, Sanhes L, Schmidt-Tanguy A, Bubenheim M, Houot R, Diouf M, Marolleau JP, Bene MC, Martin A, Lamy T. Results from a prospective, open-label, phase II trial of bendamustine in refractory or relapsed T-cell lymphomas: the BENTLY trial. J Clin Oncol. 2013 Jan 1;31(1):104-10. doi: 10.1200/JCO.2012.43.7285. Epub 2012 Oct 29. PMID 23109692